CLINICAL TRIAL: NCT03264352
Title: Intervention for High-normal Blood Pressure in Adults With Type 2 Diabetes
Acronym: IPAD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: XueQing Yu (Other)
Responsible Party: Sponsor-Investigator, XueQing Yu, Director of the Guangdong Provincial People's Hospital, Guangdong Provincial People's Hospital
Organization: Guangdong Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GDREC2017192H
Record Dates: First submitted 2017-08-21; First posted 2017-08-29 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2; Adverse Event; Blood Pressure; Prehypertension; Cardiovascular Risk Factor
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prehypertension | interventions — allisartan isoproxil; Amlodipine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intensive treatment group (Active Comparator): Real antihypertensive agents will be provided for this arm, to decrease systolic BP to lower than 120 mm Hg. In this group, the following study medications will be used: tablets with Allisartan Isoproxil 240 mg (first-line medication); tablets with Amlodipine 5 mg (second-line medication). Treatment will be started with Allisartan 240 mg. If necessary to reach the BP goal, Amlodipine (first 5 mg or then 10 mg daily) will be given in addition. If intolerable side effects occur, first-line medication may be replaced by second-line medication.
  Interventions: Drug: Allisartan Isoproxil; Drug: Amlodipine 5mg
- standard treatment group (Placebo Comparator): In this arm participants are followed up and no medications be used until BP becomes ≥ 140 mm Hg systolic and/or 90 mm Hg diastolic. Medications are determined by investigators in lines with recommendations by current Chinese guidelines to decrease BP to lower than 140 mm Hg systolic and to lower than 90 mm Hg diastolic.
  Interventions: Other: Standard treatment by current guideline

INTERVENTIONS:
Drug: Allisartan Isoproxil — Allisartan Isoproxil 240mg daily will be used to lower BP to below 120 mm Hg systolic.
  Other Names: Xinlitan
  Arms: intensive treatment group
Drug: Amlodipine 5mg — Amlodipine 5mg daily will be added to Allisartan Isoproxil and afterwards increased to 10mg daily, if necessary to reach the blood pressure goal (below 120 mm Hg systolic).
  Other Names: Qiaohean
  Arms: intensive treatment group
Other: Standard treatment by current guideline — No BP-lowering medications are used until BP becomes ≥ 140 mm Hg systolic and/or 90 mm Hg diastolic. Medications are determined by investigators in lines with recommendations by current Chinese guidelines to decrease BP to lower than 140 mm Hg systolic and to lower than 90 mm Hg diastolic.
  Arms: standard treatment group

SUMMARY:
Lowering of blood pressure (BP) in high-risk hypertensive individuals reduces major adverse cardiovascular and cerebrovascular events. Diabetic patients with hypertension benefit from BP lowering treatment. The present trial, IPAD in brief, is a randomized, open-label, parallel-designed, multicenter study involving nearly 12,000 patients to be recruited and to be followed up for a median of four years. IPAD tests the hypothesis that antihypertensive medications in adults with type 2 diabetes, whose seated BP 120-139 mm Hg systolic and below 90 mm Hg diastolic, results in 20% difference in the incidence of major adverse cardiovascular and cerebrovascular events. During follow-up for participants in the intensive group, the sitting systolic pressure should be decreased to below 120 mm Hg, by titration and combination of the study medications of an angiotensin type-1 receptor blocker Allisartan (240 mg/day), a dihydropyridine calcium-channel blocker (amlodipine 5-10 mg/day), and/or other medications if necessary. For those in the standard group, the sitting systolic pressure should be monitored and controlled below 140 mm Hg.

DETAILED DESCRIPTION:
The IPAD trial is a randomized, open-label, parallel-designed, multicenter study. 11,414 patients will be recruited in three years with a median follow up of four years. IPAD tests the hypothesis that intensive antihypertensive medical therapy in adult patients with type 2 diabetes, whose seated BP ranges from 120 to 139 mm Hg systolic and < 90 mm Hg diastolic, results in 20% reduction in the incidence of major adverse cardiovascular and cerebrovascular events (the primary endpoint), a composite of stroke, cardiovascular death, nonfatal myocardial infarction (MI), hospitalization for heart failure (HF) and hospitalization for unstable angina. Secondary endpoints of this study include: stroke; cardiovascular death; MI; hospitalization for HF; hospitalization for unstable angina; all-cause mortality; overt albuminuria; worsened renal function (the estimated glomerular filtration rate decreased by > 30% from baseline); end-stage renal disease; development of diabetic retinopathy that needs interventional operation; peripheral arterial diseases; new on-set atrial fibrillation or flutter; cancer; decline of health-related quality of life. Inclusion criteria for the study include T2DM patients aged between 45 and 79 years within the aforementioned BP ranges. for participants in the intensive group, the sitting systolic BP should decrease to < 120 mm Hg, using titration and combination of study medications consisting of an angiotensin type-1 receptor blocker Allisartan (240 mg/day) and a dihydropyridine calcium-channel blocker (amlodipine 5-10 mg/day), and/or other medications if necessary.For those in the standard group, the sitting systolic pressure should be monitored and controlled below 140 mm Hg. Across the whole study, 820 primary endpoints are expected to occur. Interim analyses will be carried out on an intention-to-treat basis. At the completion of the trial, both an intention-to-treat and a per-protocol analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* irrespective of sex;
* aged between 45 and 79 years;
* with office-measured seated BP 120-139 mm Hg systolic and below 90 mm Hg diastolic;
* diagnosed of type 2 diabetes mellitus (T2DM), currently on diabetic therapy;
* informed consent provided and long-term follow-up possible

Exclusion Criteria:

* poor control of blood glucose, HbA1c > 10.0%
* administration of any antihypertensive medications within 1 month;
* a history of hypoglycemic coma / seizure;
* confirmed diagnosis of type 1 diabetes mellitus;
* alanine-aminotransferase (ALT) or aspartate-aminotransferase (AST) over three times the upper limit of normal;
* estimated glomerular filtration rate < 45 ml/min/1.73m2;
* a history of congestive heart failure with left ventricular ejection fraction < 40%;
* coronary artery disease requiring RAS blockers for secondary prevention;
* acute on-set of stroke within 6 months prior to randomization;
* a ratio of urinary albumin (in mg/L) to urinary creatinine (in g/L) (ACR) ≥ 300 mg/g;
* known contraindications for the active study medications;
* a history of psychological or mental disorder;
* pregnancy or currently planning to have babies or lactation;
* severe diseases such as severe heart diseases;
* an expected residual life span less than 3 years;
* a malignancy that clinical investigators consider as unsuitable to participate;
* currently participating in another clinical trial.

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11414 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Composite of Major Adverse Cardiovascular and Cerebrovascular Events | From date of randomization until the date of first documented incidence of the major adverse cardiovascular events prespecified, whichever comes first, assessed up to 60 months
  The major adverse cardiovascular and cerebrovascular events defined in the study include cardiovascular death, nonfatal stroke, nonfatal myocardial infarction, hospitalization for congestive heart failure and hospitalization for unstable angina.

SECONDARY OUTCOMES:
Stroke | From date of randomization until the date of first documented incidence of stroke, assessed up to 60 months.
  Stroke (ICD-Code I60, I61, I63, I64) is a focal neurological deficit with symptoms continuing for more than 24 hours or leading to death with no apparent cause other than vascular. Stroke as an endpoint in IPAD includes definite ischemic stroke, primary intracerebral hemorrhage and subarachnoid hemorrhage with evidence from CT or MRI scan within 14 days of onset or autopsy confirmation, and stroke of unknown type etiology when CT, MRI, or autopsy are not done and information is inadequate to diagnose the etiology definitely.
Cardiovascular Death | From date of randomization until the date of cardiovascular death, assessed up to 60 months.
  Cardiovascular death include death caused by stroke, MI, HF, sudden death or any other death attributed to cardiovascular diseases. Sudden death (ICD-Code I46.1, R96) encompasses any death of unknown origin occurring instantly or within an estimated 24 hours after the onset of acute symptoms as well as unattended death for which no likely cause can be established by autopsy or recent medical history.
Acute Myocardial Infarction | From date of randomization until the date of first documented incidence of acute MI, assessed up to 60 months.
  Acute myocardial infarction (MI) (ICD-Code I21) is defined when any one of the following criteria occurs. (1) Detection of a rise and/or fall of cardiac biomarker values, with at least one value above the 99th percentile upper reference limit and with at least one of the following manifestations: symptoms of ischaemia that should have lasted for at least 30 minutes and should not have been responsive to sublingual administration of nitrates; new or presumed new significant ST-segment-T wave changes or new left bundle branch block (LBBB); development of pathological Q waves in the ECG; imaging evidence of new loss of viable myocardium or new regional wall motion abnormality. (2) Identification of an intracoronary thrombus by angiography or autopsy. (3) Cardiac death with symptoms suggestive of myocardial ischaemia and presumed new ischaemic ECG changes or new LBBB, but death occurred before cardiac biomarkers were obtained, or before cardiac biomarker values would be increased.
Hospitalization of Unstable Angina | From date of randomization until the date of first documented hospitalization of unstable angina, assessed up to 60 months.
  Unstable angina (ICD-Code I20.0) is defined as new onset or worsening angina pectoris requiring hospitalization with angiographically documented coronary atherosclerosis or transient electrocardiographic changes of the ST-segment or T-wave without evidence for myocardial necrosis. This diagnosis excludes patients with angina pectoris admitted to the hospital only for investigation.
Hospitalization of Congestive Heart Failure | From date of randomization until the date of first documented hospitalization of HF, assessed up to 60 months.
  Congestive heart failure (HF) (ICD-Code I50) requires the presence of three conditions, namely symptoms, such as dyspnea, clinical signs, such as ankle edema or crepitations, and the necessity to initiate treatment with open-label diuretics, vasodilators or antihypertensive drugs. HF cases may also be adjudicated as chronic stable HF but this is not considered an outcome of the present study.
All-cause Mortality | From date of randomization until the date of death from any causes, assessed up to 60 months.
  All-cause mortality refers to death from any causes.
Overt Albuminuria | From date of randomization until the date of confirmed development of overt albuminuria, assessed up to 60 months.
  Overt albuminuria is defined as a ratio of urinary albumin (in mg/L) to urinary creatinine (in g/L) in urine specimens of at least 300 mg/g.
Worsened Renal Function | From date of randomization until the date of first documented incidence of this event, assessed up to 60 months.
  Estimated glomerular filtration rate (eGFR) decreased by more than 30% as compared with baseline
End-Stage Renal Disease | From date of randomization until the date of documented diagnosis of end-stage renal disease, assessed up to 60 months.
  End-stage renal disease (ICD-Code N18.5) is the need for long-term renal replacement therapy (dialysis).
Diabetic Retinopathy Requiring Interventional Operation or Surgery | From date of randomization until the date of first documented interventional or surgical operation for diabetic retinopathy, assessed up to 60 months.
  Diabetic retinopathy requiring interventional operation or surgery is defined as the confirmed diagnosis of diabetic retinopathy, indicated for interventional operation or surgery, which is documented by ophthalmologists.
Peripheral Arterial Diseases Requiring Revascularization | From date of randomization until the date of first documented revascularization for peripheral arterial diseases, assessed up to 60 months.
  Peripheral arterial diseases requiring revascularization are defined as the confirmed diagnosis of any one of the peripheral arterial diseases indicated for revascularization.
New Atrial Fibrillation or Flutter | From date of randomization until the date of first documented incidence of atrial fibrillation or flutter, assessed up to 60 months.
  Atrial fibrillation or flutter is confirmed and documented with electrocardiogram indicating the occurence of atrial fibrillation or flutter. New development of atrial fibrillation or flutter is defined only if a participant at baseline has no history of and his or her electrocardiogram shows no signs of atrial fibrillation or flutter.
Decline of Health-related Quality of Life | up to 60 months
  Decline of Health-related Quality of Life, which is assessed using the EQ-5D-5L QOL questionnaire.
Cancer | From date of randomization until the date of first confirmed diagnosis of a cancer of any type, assessed up to 60 months.
  Cancer defined in the present study is recorded only when there is pathologically confirmed evidence.

CONTACTS AND LOCATIONS:
Overall Officials: Jiyan Chen, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China